CLINICAL TRIAL: NCT02659358
Title: The Biosensor Study: Exploratory Study Evaluating the Use of Wearable Biosensors and Patient Reported Outcomes (PROs) to Assess Performance Status and Distress in Patients With Cancer
Brief Title: Evaluating the Use of Wearable Biosensors and PROs to Assess Performance Status in Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Arvind Shinde, Faculty Physician, Cedars-Sinai Medical Center
Other Study IDs: IIT2015-10-Shinde-Biosens
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Neoplasms
Keywords: Advanced solid malignancy; Activity monitor; Biosensor; Fitbit; Patient Reported Outcomes (PRO); Stage 3/4 cancer; Performance Status; Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
MeSH Terms: conditions — Neoplasms | interventions — Biosensing Techniques; Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biosensor + Patient Reported Outcomes (PRO): Participants will wear a biosensor (Fitbit Charge HR®) continuously for a period of 15 days and respond to PROMIS questionnaires. This is not a chemotherapy or treatment-intervention trial.
  Interventions: Device: Fitbit Charge HR®

INTERVENTIONS:
Device: Fitbit Charge HR® — A wrist worn biosensor, the Fitbit Charge HR® has sensor capability, good battery life, water resistant, Bluetooth capabilities, and provides accessible data.
  Other Names: Biosensor; Activity monitor

SUMMARY:
The purpose of this study is to evaluate the association between wearable biosensor data, performance status and patient-reported outcomes in cancer patients. Participants in this study will wear a biosensor (Fitbit Charge HR®) for 15 days and respond to questionnaires that will assess patient reported outcome measures including physical function, emotional distress, pain interference, sleep disturbance and fatigue.

Eligible patients will have a diagnosis of advanced cancer. Patients must be greater than 18 years of age and be English speaking due to the questionnaires that will be administered during the study. Patients must also be ambulatory (use of walking aids, such as cane and rollator, is acceptable) and have access to a smartphone with internet access (IOS or Android). It is also necessary for patients to have scheduled oncology clinic visits at least once every 2 weeks.

DETAILED DESCRIPTION:
This study aims to measure association between biosensor data, performance status and patient-reported outcomes. This study will also evaluate the feasibility of using Fitbit activity monitors in a cancer population to capture objective activity data. The study will be recruiting patients with advanced cancer diagnoses (stage 3 or 4) and will be referred by the treating oncologist. This is an exploratory study that will follow patients with stage 3-4 cancer for a period of 15 days. Subjects will be provided with a Fitbt Charge HR® activity monitor. They will be requested to wear the Fitbit Charge HR® at all times, except for while bathing or performing other activities where the activity monitor can become submerged in water. Subjects will be asked to wear the Fitbit Charge HR® for two weeks. They will be seen in the clinic at baseline, at the end of week 1 (day 8) and at end of 2 weeks (day 15) for physical exam, evaluation of performance status by both treating oncologist and practice nurse using standardized scales and administration of PROMIS® questionnaires. Patients will be followed up to 6 months after the last clinic visit for adverse events, hospitalization and survival. Thirty subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced solid malignancy (Stage 3 or 4) with measurable disease, who are being followed by an oncologist
* 18 years or older
* English speaking
* Ambulatory (use of walking aids, such as cane and rollator, is acceptable)
* Access to IOS or Android smartphone with internet access
* Expected to have oncology clinic visits at least once every 2 weeks
* Have an understanding, ability, and willingness to fully comply with study procedures and restrictions
* Ability to consent

Exclusion Criteria:

* Allergy to surgical steel or elastomer/rubber
* Using a pacemaker, implantable cardiac defibrillator, neurostimulator, hearing aids, cochlear implants, or other electronic medical equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01-24 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Physical activity as measured using Fitbit Charge HR (composite of mean daily steps and stairs per day, mean resting heart rate, mean daily active minutes and time sedentary, stairs climbed) | 15 days
  Data will be compared to reference standards to answer primary objective.
Performance status as measured with with Eastern Cooperative Oncology Group performance status (ECOG-PS) scale | 15 days
  ECOG PS will be compared to physical activity as measured using biosensor data (Outcome 1)
Performance status as measured with Karnofsky Performance Status (KPS) | 15 days
  KPS will be compared to physical activity as measured using biosensor data (Outcome 1)
Patient-reported physical function summary using NIH Patient Reported Outcome Measurement System (PROMIS®) tool | 15 days
  Mean weekly summary score of physical function from NIH PROMIS® tools will be compared to biosensor metrics (outcome 1) and performance status (Outcomes 2 and 3)

SECONDARY OUTCOMES:
Summary score of emotional distress as measured using NIH PROMIS® questionnaire | 15 days
Summary score of pain interference as measured using NIH PROMIS® questionnaire | 15 days
Summary score of fatigue as measured using NIH PROMIS® questionnaire | 15 days
Summary score of sleep interference as measured using NIH PROMIS® questionnaire | 15 days
Presence of frailty phenotype | 15 days
  Using Fried's definition, frailty is present if ≥3 characteristics of frailty are present. Association between measures of frailty and biosensor data will be measured.
Feasibility defined as proportion of time Fitbit is worn during study period (4 of 7 days worn in the study) | 15 days
  This will be measured by using the duration of time that the Fitbit Charge HR is worn and recording data during the study. Recorded data from the device for 4 of each 7 days of the study (at least 16 hrs of each day) will support feasibility of utilizing the Fitbit Charge HR to collect data. Feasibility of collecting PROMIS® tool responses will be determined by percentage of completed PROMIS® tools. PROMIS® tool completion rates of >50% will support the feasibility of current method of utilizing PROMIS® tools to collect PROs.
Occurrence of any chemotoxicity (using CTCAE v4) within patients who are undergoing treatment for their condition during time of study | 4 weeks after completion of study
  Patients enrolling in the study will be treated for their condition (per standard of care). We will capture the occurrence of toxicities form their respective treatments to determine how physical activity (as measured using the biosensor) predicts the events.
Occurrence of hospitalization (yes/no) | At 3 and 6 months after completion of 15 day study
  Will follow-up with patients at specified time points to determine whether the patient experienced any hospitalizations (binary event) to determine whether baseline activity levels (as measured using biosensor) predicts the event.
Number of hospitalizations | At 3 and 6 months after completion of 15 day study
  Will follow-up with patients at specified time points to determine how many hospitalizations the patient experienced (continuous) to evaluate whether baseline activity levels (as measured using biosensor) predicts the number of hospitalizations.
Mortality | At 3 and 6 months after completion of 15 day study
  Determine whether baseline activity levels as measured using biosensor predict occurrence of death within the specified time frame

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Shinde, MD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No